CLINICAL TRIAL: NCT01833845
Title: An Open-Label Study to Evaluate the Efficacy, Safety and Tolerability of Ribavirin Monotherapy Followed by Combined Treatment With Ribavirin and Hydroxychloroquine in Patients Infected With Hepatitis C
Brief Title: Efficacy, Safety and Tolerability of Ribavirin Monotherapy Followed by Combined Treatment With Ribavirin and Hydroxychloroquine in Patients Infected With Hepatitis C
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: due to failure to recruit subjects
Sponsor: BioLineRx, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BL-8020.01
Record Dates: First submitted 2013-04-15; First posted 2013-04-17 (Estimated); Results first posted 2014-08-28 (Estimated); Last update posted 2014-08-28 (Estimated); Status verified 2014-08

CONDITIONS: Hepatitis C
Keywords: HCV; Hepatitis C; Hep-C
MeSH Terms: conditions — Hepatitis C | interventions — Ribavirin; Hydroxychloroquine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ribavirin+HCQ (Experimental): Administration of RBV monotherapy for a period of 8 weeks following administration of up to 16 weeks combination therapy with ribavirin(RBV) plus Hydroxychloroquine(HCQ).
  Interventions: Drug: Ribavirin; Drug: Hydroxychloroquine

INTERVENTIONS:
Drug: Ribavirin — weight-based doses (1000 mg/day administered BID [twice daily] for subjects ≤ 75 kg and 1200 mg/day administered BID for subjects > 75 kg). Those subjects receiving 1000 mg/day RBV will take 2 tablets of 200 mg/tablet in the morning and 3 tablets in the evening, and those subjects receiving 1200 mg/day RBV will take 3 tablets morning and evening.
  Other Names: RBV
Drug: Hydroxychloroquine — subjects will receive HCQ 575 mg administered as a single tablet once daily (QD)
  Other Names: HCQ

SUMMARY:
Proof-of Concept, Open-Label, Two-Stage Study without Direct Individual Benefit The proposed study design consists of two treatment periods and one treatment arm. Treatment Period 1 involves the administration of RBV monotherapy for a period of 8 weeks and Treatment Period 2 involves administration of up to 16 weeks combination therapy with RBV plus HCQ.

DETAILED DESCRIPTION:
Patients who provide their informed consent and conform to all the inclusion and none of the exclusion criteria will be enrolled into the study and will receive RBV monotherapy for 8 weeks. Subjects will receive weight-based doses (1000 mg/day administered BID [twice daily] for subjects ≤ 75 kg and 1200 mg/day administered BID for subjects > 75 kg). Those subjects receiving 1000 mg/day RBV will take 2 tablets of 200 mg/tablet in the morning and 3 tablets in the evening, and those subjects receiving 1200 mg/day RBV will take 3 tablets morning and evening.

During Treatment Period 2, subjects will receive HCQ 575 mg administered as a single tablet once daily (QD), in addition to continuing the same dose of RBV that was administered during Treatment Period 1, as combination therapy for up to 16 weeks.

Subjects will undergo regular blood sampling throughout Treatment Periods 1 and 2 to measure viral response (HCV RNA). Safety will be assessed throughout the study by collection of adverse event (AE) and concomitant medication data, and routine monitoring of laboratory safety tests, vital signs and 12-lead electrocardiograms (ECG).

Subjects will have their viral response tested following 12 weeks of combination therapy; those who show < 1 log decline in viral load during the combination therapy will have the opportunity to withdraw and transfer to standard of care (SoC) treatment following performance of the "End of Study Treatment" visit.

On completion of study treatment, subjects will be allowed to transfer immediately to SoC treatment in order to maximize the benefit of any reduced viral load resulting from combination therapy with RBV plus HCQ. Subjects will attend the clinical site for an "End of Study Treatment" visit within 2 weeks of the final dose of combination treatment with RBV plus HCQ during which they will undergo a final measurement of HCV RNA, safety assessments as described above and a full physical and ophthalmic examination. The "End of Study Treatment" visit may take place on the same day as the final study visit at week 24.

In the event of subjects achieving viral undetectability during combination therapy, the relevant subjects may be administered additional combination therapy to achieve a total of 24 weeks of viral undetectability. If combination dosing with RBV plus HCQ continues for more than 16 weeks, subjects will continue to attend the clinical site and undergo assessment of safety and viral load at the discretion of the Investigator. However, treatment beyond 16 weeks of combination therapy will be considered compassionate use and will not be considered part of the study. In these subjects, the "End of Study Treatment" visit will take place no more than 2 weeks after the Week 24 visit.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, age ≥ 18.
2. Subjects diagnosed to have positive HCV antibodies.
3. Subject is diagnosed to have detectable HCV RNA by PCR.
4. FibroTest or FibroScan or liver biopsy showing a METAVIR score ≤ F2 and/or

   ≤ A2 within 2 years of the screening visit.
5. Subject is a non-responder (null or partial ) OR relapsed following prior Peg-IFN and RBV based treatment lasting for at least 12 consecutive weeks.
6. Platelet count greater than or equal to 100,000 cells/mm3.
7. Absolute neutrophil count (ANC) greater than or equal to 1500 cells/mm3.
8. Subjects able to comprehend and give written informed consent for participation in this study.
9. Women of childbearing potential and all men must agree to use an approved form of contraception (e.g., oral, transdermal patch, implanted contraceptives, intrauterine device, diaphragm, condom, abstinence or surgical sterility) prior to study entry and for the duration of study participation through 7 months after the last dose of study medication. Confirmation that the female patient is not pregnant must be established by a negative serum β-human chorionic gonadotropin (β-hCG) pregnancy test result obtained during screening. Pregnancy testing is not required for post-menopausal or surgically sterilized women.
10. Subject is willing to be treated and commit to all visits

Exclusion Criteria:

1. Contraindication or hypersensitivity to one of the study drugs (HCQ or RBV).
2. Patient has anemia (male <13 g/dL; female <12 g/dL), elevated ALT and/or AST >10 x ULN or elevated creatinine (>1.5 mg/dL).
3. Concomitant liver disease other than hepatitis C: alcoholic liver disease, autoimmune hepatitis, Wilson's disease, hemochromatosis, alpha-1 antitrypsin deficiency.
4. Decompensated cirrhosis (Child Pugh >A).
5. Ongoing hepatocellular carcinoma (suggestive imaging study or alpha-fetoprotein (AFP) >50 ng/mL).
6. Hepatitis B or Human Immunodeficiency Virus (HIV1 or HIV2) co-infection.
7. Clinically relevant ECG abnormalities on screening or baseline 12-lead ECG, e.g.,

   * QTc interval (QTcB or QTcF > 450 ms in males and > 470 ms in females);
   * Notable resting bradycardia (HR < 40 bpm);
   * Any other significant abnormality suggestive of structural heart disease.
8. Family history of congenital long QT syndrome.
9. Clinically significant abnormalities on ophthalmic examination.
10. Major uncontrolled psychiatric illness. Minor or situational depressions are allowed.
11. History of hemoglobinopathy (e.g., thalassemia) or any other cause of or tendency to hemolysis (e.g., G-6-PD deficiency).
12. Active illicit drug or alcohol abuse.
13. Serious co-morbid conditions such as: heart failure, significant coronary heart disease, chronic obstructive pulmonary disease, poorly controlled diabetes, autoimmune disorders and any malignant diseases (except in situ carcinomas or basal cell carcinoma) in the previous 5 years.
14. Patients with chronic renal insufficiency, creatinine clearance < 50 mL/minute and/or undergoing haemodialysis.
15. Patients with porphyria or psoriasis.
16. Ongoing concomitant treatment with azathioprine, digoxin or medications known to prolong QT interval.
17. History of organ transplantation.
18. Pregnancy, breast-feeding or unwillingness to practice double contraception or abstinence by the subject of childbearing potential or partner.
19. Concurrent participation in any other clinical study or within 180 days 20.Patients with inability to communicate well with the Investigators and staff (i.e., language problem, poor mental development or impaired cerebral function) or any other condition that in the opinion of the Investigator will place the patient at risk or prevent protocol compliance.

    -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2013-04; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stanislas Pol, MD, Principal Investigator — Cochin Hospital; Marc Bourliere, MD, Principal Investigator — S.Joseph Hospital
Locations (2):
- France (2):
  - Hospital St. Joseph, Marseille
  - Cochin Hospital, Paris

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ribavirin+HCQ
Started | 4
Completed | 4
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: 40 subjects were planned to be included in the study; however, due to the Sponsor's decision, the study was terminated prematurely after 4 subjects had completed the study, due to failure to recruit subjects
Arm/Group | Ribavirin+HCQ
Number analyzed (Participants) | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.8 (6.0)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 3
Region of Enrollment [Number; unit: participants]
  France | 4

OUTCOME MEASURES:

1. Primary Outcome: Efficacy
Description: To evaluate the effect of 16-week combination therapy with RBV plus HCQ following 8 weeks of monotherapy with RBV in HCV-infected patients.
Time Frame: 24 weeks
Reporting Status: Not Posted

2. Primary Outcome: Safety: Number of Participants With Adverse Events
Description: Safety was assessed throughout study by collection of adverse event and concomitant medication data, and routine monitoring of lab safety tests, physical exams, ophthalmic examination, vital signs and 12 lead electrocardiograms.
Time Frame: all 24 weeks
Measure: Number; unit: participants
Arm/Group | Ribavirin+HCQ
Number analyzed (Participants) | 4
participants | 4

3. Secondary Outcome: Efficacy
Description: To evaluate the efficacy of 8 weeks monotherapy with RBV in HCV-infected patients.
Time Frame: 8 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Ribavirin+HCQ
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 4/4
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ribavirin+HCQ (N=4)
Upper abdominal pain (Gastrointestinal disorders) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Dysgeusia (Nervous system disorders) | 1 (1)
Asthenia (Gastrointestinal disorders) | 2 (2)
insomnia (Psychiatric disorders) | 2 (2)
dry eye (Eye disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The publication of the results of the Research in their entirety or in part, will be at the sole initiative of BIOLINERX Ltd. Reference to the results of the search cannot be made without the prior written agreement of BioLineRx Ltd..